CLINICAL TRIAL: NCT06503939
Title: Etiology Analysis of Chronic Cough After COVID-19 Infection and Research on the Efficacy of ICS or ICS/LABA
Status: Enrolling by invitation | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: Z-2017-24-2301
Record Dates: First submitted 2024-07-14; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Cough
Keywords: COVID-19
MeSH Terms: conditions — Chronic Cough; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study collected 600 patients, evaluated whether patients had airway hyperreactivity, airway inflammation, specific types and allergic reactions, comprehensively analyzed and classified the causes of chronic cough in patients, and evaluated and compared the improvement of cough symptoms and quality of life after ICS or ICS/LABA treatment.

DETAILED DESCRIPTION:
The subjects of this study were patients with chronic cough who were admitted to the Department of Respiratory and Critical Care Medicine, Xiangya Hospital, Central South University from September 1, 2023 to December 31, 2024. Patients are registered if they meet all of the following criteria: (1) ≥18 years of age; (2) A clear history of COVID-19 infection with a positive nucleic acid or antigen test before chronic cough;(3) Persistent cough for more than 8 weeks after the acute phase of COVID-19 infection has disappeared; (4) Chest X-ray and/or chest CT without significant evidence of lung disease; (5) No history of chronic cough (>8 weeks) prior to COVID-19 infection. Patients who met any of the following criteria were excluded: (1) Patients refused pulmonary function, blood tests; (2) The patient has previously been diagnosed with respiratory diseases with cough as one of the main symptoms, including cough variant asthma, allergic bronchitis, eosinophilic bronchitis, gastroesophageal reflux disease, chronic obstructive pulmonary disease, chronic bronchitis, bronchiectasis, interstitial lung disease, pulmonary/tracheobronchial tuberculosis, etc.; (3) Patients who are pregnant or breastfeeding; (4) The patient's medical records are incomplete; (5) Patients lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. A clear history of COVID-19 infection with a positive nucleic acid or antigen test before chronic cough;
3. Persistent cough for more than 8 weeks after the acute phase of COVID-19 infection has disappeared;
4. Chest X-ray and/or chest CT without significant evidence of lung disease;
5. No history of chronic cough (>8 weeks) prior to COVID-19 infection.

Exclusion Criteria:

1. The patient refused pulmonary function and blood tests;
2. The patient has previously been diagnosed with respiratory diseases with cough as one of the main symptoms, including cough variant asthma, allergic bronchitis, eosinophilic bronchitis, gastroesophageal reflux disease, chronic obstructive pulmonary disease, chronic bronchitis, bronchiectasis, interstitial lung disease, pulmonary/tracheobronchial tuberculosis, etc.;
3. Patients who are pregnant or breastfeeding;
4. The patient's medical records are incomplete;
5. Patients lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons who meet the above inclusion criteria and for whom no exclusion criteria exist
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The etiology of chronic cough was comprehensively analyzed and classified. | 2023.09-2024.12

SECONDARY OUTCOMES:
To evaluate and compare cough symptoms and quality of life improvement after ICS or ICS/LABA treatment. | 2023.09-2024.12

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jiang, Doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China